CLINICAL TRIAL: NCT05827913
Title: Evaluation of the Efficacy and Safety of Polylevolactic Acid Injection Filling Combined With 1565nm Non-ablative Fractional Laser in the Treatment of Striae Distensae
Brief Title: Efficacy and Safety of Polylevolactic Acid Injection Combined With 1565nm Non-ablative Fractional Laser in the Treatment of Striae Distensae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: XijingH-PF-KY20232083
Record Dates: First submitted 2023-03-29; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-03

CONDITIONS: Striae Distensae
Keywords: Polylevolactic Acid; Striae Distensae; 1565nm Non-ablative Fractional Laser; treatment
MeSH Terms: conditions — Striae Distensae

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Polylevolactic Acid Injection (Experimental): Polylevolactic Acid Injection in SD
  Interventions: Device: Polylevolactic Acid Injection
- Fractional Laser (Active Comparator): 1565nm Non-ablative Fractional Laser treatment in SD
  Interventions: Device: 1565nm Non-ablative Fractional Laser
- combination treatment (Active Comparator): Polylevolactic Acid injection combined with 1565nm Non-ablative Fractional Laser treatment in SD
  Interventions: Device: Polylevolactic Acid Injection combined with 1565nm Non-ablative Fractional Laser

INTERVENTIONS:
Device: Polylevolactic Acid Injection — The patient was placed in a flat recumbent position and subjected to topical anesthesia with lidocaine cream for those who were unable to tolerate pain. According to the location and degree of indentation of the atrophic stria, a conventional disinfection towel is placed and injected into the subcutaneous and deep dermis. Use left thumb and index finger to press or tighten the skin from both sides to the middle. Depending on the location of the SD, determine the injection direction. During linear injection, the injection starts from the distal end of the SD, and then the injection is withdrawn until the SD subsides. Apply uniform force and withdraw the needle at a uniform speed. Stop the injection before the needle is pulled out of the skin, To avoid too shallow an injection.
  Arms: Polylevolactic Acid Injection
Device: 1565nm Non-ablative Fractional Laser — M22-ResurFx laser (Lumenis Medical Company, USA) was used for treatment, with a wavelength of 1565 nm, a selected energy of 45 mJ, and a lattice density of 200 dots/cm2. The end point reaction was erythema and wind masses at the treatment site.
  Arms: Fractional Laser
Device: Polylevolactic Acid Injection combined with 1565nm Non-ablative Fractional Laser — combination of the two treatments described above
  Arms: combination treatment

SUMMARY:
1. Striae distensae (SD), also known as stretch marks, are common, permanent dermal lesions that can be symptomatic and are considered aesthetically undesirable; thus, they pose a significant psychosocial and therapeutic challenge. SD arise in areas of dermal stretching and most commonly occur on the abdomen, breasts, buttocks, and thighs. Most literature has described SD during pregnancy(striae gravidarum) and puberty, with reported prevalences varying from 11% to 88%. Hormonal influences, reduced genetic expression of fibronectin, collagen, and elastin, and mechanical stretching of the skin have all been postulated to contribute to SD formation. In the acute phase, SD appear as red/violaceous lesions (striae rubrae; SR) that can be raised and symptomatic. The chronic form (striae albae; SA) exists as hypopigmented dermal depressions.
2. Polylevolactic Acid(PLLA) is at present one of the most promising biodegradable polymers (biopolymers) and has been the subject of abundant literature over the last decade. PLLA can be processed with a large number of techniques and is commercially available (large-scale production) in a wide range of grades.
3. Previous studies have found that 1565-nm laser can promote the synthesis of types I, III, and VII collagen and elastin, as well as the remodeling of dermal collagen. According to previous studies, dermal collagen deposition and remodeling may be related to the mechanism by which 1565-nm laser improves SD.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-50 years old, regardless of gender;
2. The clinical diagnosis was atrophic stria;
3. Patients with normal blood routine, liver and kidney function, and preoperative infection;
4. Able to communicate well with researchers and comply with the overall test requirements;
5. Willing to take and retain photos before and after treatment;
6. Volunteer and sign an informed consent form.

Exclusion Criteria:

1. Scar constitution;
2. Acute or chronic skin infections (including bacteria, viruses, and fungi) exist near the treatment area;
3. Those who are allergic to any component of the product;
4. Those who have been injected with anticoagulant drugs;
5. Those who have used other drugs, other substances, and other implant agents;
6. Patients with severe primary and psychiatric disorders such as heart, brain, liver, kidney, hematopoietic system, endocrine system, etc;
7. History of peripheral vascular disease, long-term alcoholism, diabetes, immunosuppression, disorder, drug abuse, etc;
8. Pregnant and lactating women;
9. Those who are critically ill and difficult to accurately evaluate the effectiveness and safety of the product.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
The treatment effect is judged by color, area, concavity and convexity, and skin elasticity | 4months
  * Color: Ranked in order as follows: Purple red pink skin color, no change 0 point, 1 point added for each shade subtracted;
    * Area: 0 point: no change, 1 point: slightly improved, 2 points: significantly improved, 3 points: basically invisible;
      * Bump sensation: 0 point: no change, 1 point: slightly improved, 2 points: significantly improved, 3 points: bump basically eliminated;
        * Skin elasticity: 0 point: no change, 1 point: slightly improved, 2 points: significantly improved, 3 points: very satisfied;
  The total score of 6-12 points is basically cured; A total score of 3-5 points is significant; Effective with a total score of 1-2; A total score ≤ 1 is invalid.
  Total effective rate of treatment=(basically cured+significantly effective+effective)/total number of cases × 100%.
  Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Prof, Principal Investigator — Dermatology Department of Xijing Hospital
Locations (1):
- Dermatology Derpartment of Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Qu H, Wang L, Xin W, Lu M, Jing H, Wang G, Gao L. Clinical Efficacy Comparisons Between Poly-L-Lactic Acid Injections and Non-Ablative 1565-nm Fractional Laser for Treatment of Striae Distensae-A Randomized Trial. J Cosmet Dermatol. 2025 Jul;24(7):e70338. doi: 10.1111/jocd.70338. PMID 40662320